CLINICAL TRIAL: NCT01843023
Title: Health Services Research: Extended Release Naltrexone for Opioid-Dependent Youth
Brief Title: Extended Release Naltrexone for Opioid-Dependent Youth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA033391-01A1 (NIH); R01DA033391 (NIH)
Record Dates: First submitted 2013-04-25; First posted 2013-04-30 (Estimated); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Drug Dependence
Keywords: opioid dependence
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders | interventions — vivitrol; Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended Release Naltrexone (Experimental): Participants randomly assigned to XR-NTX who do not have opioid withdrawal signs or symptoms within 4 hours of administration of the 25 mg oral dose naltrexone will be given an intramuscular injection of XR-NTX [Vivitrol®] at a dose of 4cc (380mg of naltrexone)] and will subsequently have the same dose administered to alternating sides of the buttocks every four weeks for up to 6 months. All participants will also receive psychosocial treatment.
  Interventions: Drug: Extended Release Naltrexone; Behavioral: Psychosocial Treatment
- Treatment as Usual (Active Comparator): Participants randomly assigned to TAU will participate in the standard youth opioid program at the treatment center which includes either buprenorphine taper or ongoing buprenorphine treatment during the 6 months of the study for as long as they and their physicians think is appropriate. The general target dose will be 12-20 mg buprenorphine per day. All participants in TAU will receive psychosocial treatment.
  Interventions: Behavioral: Psychosocial Treatment; Drug: Buprenorphine

INTERVENTIONS:
Drug: Extended Release Naltrexone — naltrexone for extended release injectable suspension
  Other Names: Vivitrol
  Arms: Extended Release Naltrexone
Behavioral: Psychosocial Treatment — Psychosocial treatment will consist of group and individual drug abuse counseling at MMTC and in the community.
Drug: Buprenorphine — Participants assigned to TAU will receive buprenorphine for opioid withdrawal and will either be tapered off the medication or will remain on it for individualized lengths of time during the six month study.
  Other Names: Suboxone; Subutex
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to compare 6-month treatment outcomes for 15-21 year old opioid-dependent youth receiving extended release naltrexone (XR-NTX) v. Treatment as Usual (TAU).

DETAILED DESCRIPTION:
This proposed study is a 6-month, two-group randomized clinical trial of XR-NTX v. TAU for 340 opioid-dependent youth ages 15-21. The study will be conducted at Mountain Manor Treatment Center, a community drug treatment program in Baltimore. TAU will consist of buprenorphine treatment of opioid withdrawal followed by counseling with or without continued buprenorphine.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual-IV criteria for opioid dependence, physiologic subtype;
* Within 3 days of admission to MMTC;
* Age between 15 and 21, inclusive;
* Able and willing to provide informed consent to be randomly assigned to XR- NTX or TAU; and for participants under 18 years of age, parental or guardian consent and participant assent.

Exclusion Criteria:

* Liver function test levels (Alanine Transaminase, Aspartate Transaminase) four times greater than normal;
* Unstable medical or psychiatric illness (e.g., schizophrenia) that might make participation hazardous;
* History of serious suicide attempt in the past 6 months;
* History of allergic reaction to naloxone, and/or naltrexone;
* Current chronic pain condition for which opioids are deemed necessary for ongoing care;
* blood coagulation disorder (e.g., hemophilia);
* Body Mass Index > 40;
* If female, pregnant, lactating, unwilling or unable (due to parental objection) to use FDA-approved contraceptive methods;
* meeting DSM-IV criteria for benzodiazepine dependence

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 288 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon G Mitchell, PhD, Principal Investigator — Friends Research Institute, Inc.
Locations (2):
- United States (2):
  - Friends Research Institute, Baltimore, Maryland
  - Mountain Manor Treatment Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended Release Naltrexone | Treatment as Usual
Started | 144 | 144
3 Months | 110 | 114
Completed | 111 | 109
Not Completed | 33 | 35
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 24 | 29
Not completed — Withdrawal by Subject | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Release Naltrexone | Treatment as Usual | Total
Number analyzed (Participants) | 144 | 144 | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 8 | 25
  Between 18 and 65 years | 127 | 136 | 263
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.18 (1.3) | 19.46 (1.2) | 19.32 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 67 | 133
  Male | 78 | 77 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 138 | 135 | 273
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 13 | 28
  White | 118 | 121 | 239
  More than one race | 8 | 8 | 16
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 144 | 144 | 288
Self-reported opioid use past 90 days [Mean (Standard Deviation); unit: days] | 65.71 (23.2) | 63.19 (23.5) | 64.45 (23.4)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use at 6 Month Follow-up
Description: To determine the relative effectiveness of XR-NTX compared to TAU for opioid-dependent youth in terms of opioid use at 6-months post-treatment entry.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: days
Arm/Group | Extended Release Naltrexone | Treatment as Usual
Number analyzed (Participants) | 111 | 109
days | 19.63 (2.55) | 18.42 (2.68)

2. Secondary Outcome: Treatment Retention
Description: To determine the relative effectiveness of XR-NTX compared to TAU for opioid-dependent youth in terms of days in treatment. Treatment defined as medications for OUD received in past 30 days at 6-month follow-up.
Time Frame: 6 months
Population: Participants who completed 6-month follow-up assessment with complete data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Extended Release Naltrexone | Treatment as Usual
Number analyzed (Participants) | 109 | 109
days | 5.53 (11.07) | 4.69 (10.16)
Statistical Analysis 1: Comparison: Extended Release Naltrexone vs Treatment as Usual; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = .558

3. Secondary Outcome: Monetized Healthcare Utilization
Description: The cost-effectiveness will be assessed using the Economic Form 90 to collect data on economic outcomes of health utilization at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: dollars
Arm/Group | Extended Release Naltrexone | Treatment as Usual
Number analyzed (Participants) | 140 | 142
dollars | 8136 (646.07) | 6629 (602.55)

4. Secondary Outcome: HIV Sex Risk Behaviors
Description: To examine the impact of XR-NTX on HIV sex-risk behaviors at 6 months. Past 90 days self-reported HIV sex risk behaviors on the Risk Assessment Battery (RAB). Minimum value 0; maximum value 24. Higher scores reflect endorsement of more risk behaviors (worse outcome).
Time Frame: 6 months
Population: Participants who completed 6-month follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended Release Naltrexone | Treatment as Usual
Number analyzed (Participants) | 111 | 109
score on a scale | 3.53 (2.23) | 3.42 (2.34)
Statistical Analysis 1: Comparison: Extended Release Naltrexone vs Treatment as Usual; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = .722

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Extended Release Naltrexone | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 1/144 | 0/144
Serious Adverse Events (participants affected / at risk) | 5/144 | 5/144
Other Adverse Events (participants affected / at risk) | 132/144 | 122/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Naltrexone (N=144) | Treatment as Usual (N=144)
Acute Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Amputation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mood Instability (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Epidural Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Naltrexone (N=144) | Treatment as Usual (N=144)
Chest Pain (Cardiac disorders) | 1 (1) | 7 (7)
Seizure (Endocrine disorders) | 2 (3) | 1 (1)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 11 (13) | 11 (11)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 15 (17) | 16 (18)
Vomitting (Gastrointestinal disorders) | 12 (14) | 15 (16)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Root Canal Infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hot flush (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 4 (6) | 4 (4)
Injection site erythema (General disorders) | 2 (4) | 1 (1)
Injection site mass (General disorders) | 12 (16) | 11 (14)
Injection site pain (General disorders) | 18 (26) | 14 (20)
Injection site pruritus (General disorders) | 2 (4) | 1 (1)
Injection site swelling (General disorders) | 5 (8) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 5 (5)
Pain (General disorders) | 9 (10) | 11 (12)
Dark urine (Hepatobiliary disorders) | 10 (11) | 9 (9)
Hepatitis C (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver function test (Hepatobiliary disorders) | 3 (3) | 0 (0)
Multiple Allergies (Immune system disorders) | 6 (6) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 11 (11) | 12 (13)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 17 (17)
Amputation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Athralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (8)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ligament Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (22) | 15 (17)
Tingling in arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cold stimulus headache (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 6 (6)
Epidural Hemorrage (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 28 (38) | 29 (36)
Unintended Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 23 (25) | 30 (33)
Depression (Psychiatric disorders) | 19 (20) | 23 (25)
Drug withdrawal syndrome (Psychiatric disorders) | 53 (68) | 52 (65)
Acute intoxication (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalized for observation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 34 (43) | 38 (45)
Irritability (Psychiatric disorders) | 15 (18) | 17 (18)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 6 (6) | 4 (4)
Suicidal Ideation (Psychiatric disorders) | 3 (3) | 8 (8)
Intentional Self Injury (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (11)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (13)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Formication (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (8)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Contusion (Vascular disorders) | 4 (4) | 2 (2)
Epistaxis (Vascular disorders) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
There was poor participant adherence to receiving the randomly assigned condition prior to inpatient discharge. For this reason, great caution is urged in interpreting outcomes based on study condition as assigned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT01843023/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT01843023/SAP_001.pdf